CLINICAL TRIAL: NCT05198466
Title: Electrical Stimulation Therapy for Recovery of Hospital-acquired Weakness in Critically Ill COVID-19 Patients - A Proof of Concept Randomized Controlled Trial
Brief Title: Electrical Stimulation for Critically Ill Post-Covid-19 Patients
Acronym: Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Avazzia, Inc (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-47781-B
Record Dates: First submitted 2022-01-18; First posted 2022-01-20 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Muscle Atrophy; Muscle Weakness
Keywords: Electrical Stimulation; Skin perfusion; Muscle dysfunction
MeSH Terms: conditions — COVID-19; Muscular Atrophy; Muscle Weakness | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention (IG) or control group (CG) with ratio of 1:1. The entire cohort will receive daily electrical stimulation (EE) in lower extremity (e.g. Gastrocnemius muscle) for up to 1 hour. The EE device will be functional for IG and non-functional for CG.
  Phase II will include previously hospitalized patients (n=20) who had recover from severe COVID-19 infection, but present persistent neuromuscular sequelae. This will be performed in an outpatient clinic. The time frame will be 4 weeks.
Who Masked: Participant, Care Provider
Masking Description: Devices may be active or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active E-Stim (Active Comparator): Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for 4 weeks (phase II).
  Interventions: Device: Electrical Stimulation
- Electrical Stimulation - Sham (Sham Comparator): Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for 4 weeks (phase II).
  Interventions: Device: Electrical Stimulation - Sham

INTERVENTIONS:
Device: Electrical Stimulation — Subjects will receive an active electrical stimulation device to wear for 1 hour daily for 4 weeks (phase II).
  Arms: Active E-Stim
Device: Electrical Stimulation - Sham — Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for 4 weeks (phase II).
  Arms: Electrical Stimulation - Sham

SUMMARY:
Unfortunately, hospital-acquired weakness is highly prevalent among COVID-19 hospitalized patients, who often require prolonged bed-rest or paralytics for an extended period of time in order to maintain oxygenation. Prolonged bed rest has been associated with pronounced loss of muscle mass that can exceed 10% over the 1st week, which leads to functional impairment and complications post-hospital discharge. Physical therapy and in-hospital mobility program may reduce the incident of hospital-acquired weakness, but they are often impractical for COVID-19 patients. In particular, conventional mobility programs are challenging for those who are being treated in an intensive Care Unit. The purpose of this study is to test feasibility and proof-of-concept effectiveness of daily use of lower extremity electrical stimulation (EE) therapy, as a practical solution to address lower extremity muscle deconditioning, to address chronic consequences of COVID-19 including hospital-acquired weakness.

DETAILED DESCRIPTION:
20 subjects that were hospitalized due to severe COVID-19 infection and present neuromuscular complications (i.e., hospital acquired weakness due to neuromyopathy) will be recruited after the first phase of this study is completed. Unlike Phase I (study for prevention), this is a proof of concept randomized control trial (RCT) study for recovery. The patients will be recruited from the COVID-19 Clinic at Baylor College of Medicine and will begin the study after being diagnosed with neuromyopathy due to prolonged hospitalization for COVID-19. This will be performed by a critical care and pulmonary specialist at the BCM COVID-19 Clinic. The entire cohort will receive daily electrical stimulation in lower extremity (e.g. Gastrocnemius, tibial anterior muscle) up to 1 hour to recover from Neuromyopathy complications and prolonged hospital stay. Participants will be randomized to intervention (IG) or control group (CG)). EE therapy will be provided using a bio-electric stimulation technology (BEST) platform (Tennant Biomodulator PRO®, AVAZZIA, Inc.). The EE device will be functional for IG and non-functional for CG. In addition to taking the device home to deliver electrical stimulation themselves, the patients will attend a weekly assessment at the McNair Campus for up to 4 weeks. The primary outcomes include between group difference and change from the baseline in muscle endurance, muscle strength, lower extremity tissue oxygen saturation, neuropathy, and muscle atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-19 patients who required hospitalization due to COVID-19 severe infection.
* Post-COVID-19 patients who required hospitalization and present neuromuscular sequelae due to COVID-19 severe infection.

Exclusion Criteria:

* Patient has a demand-type cardiac pacemaker, implanted defibrillator or other implanted electronic device.
* Active wound infection.
* Below the knee amputations.
* Based on the clinicians decision whether the patient is eligible for the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Zulbaran-Rojas A, Lee M, Bara RO, Flores-Camargo A, Spitz G, Finco MG, Bagheri AB, Modi D, Shaib F, Najafi B. Electrical stimulation to regain lower extremity muscle perfusion and endurance in patients with post-acute sequelae of SARS CoV-2: A randomized controlled trial. Physiol Rep. 2023 Mar;11(5):e15636. doi: 10.14814/phy2.15636. PMID 36905161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note that these results only include Post-Covid-19 Patients (Phase II).
Period: Overall Study
Arm/Group | Active E-Stim | Electrical Stimulation - Sham
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active E-Stim | Electrical Stimulation - Sham | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.10 (9.86) | 52.38 (7.44) | 51.74 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Gastrocnemius Muscle Endurance (Muscle Sustained Contraction) in Response to Electrical Stimulation
Description: Gastrocnemius muscle endurance in response to 5 minutes of electrical stimulation therapy will be assessed with surface electromyography using a validated non-invasive device (Delsys Trino Wireless EMG System, MA, US).
Time Frame: an average of 4 weeks (Phase II)
Measure: Mean (Standard Error); unit: miliVolts
Arm/Group | Active E-Stim | Electrical Stimulation - Sham
Number analyzed (Participants) | 10 | 8
miliVolts | 363.04 (1.56) | 359.55 (2.04)

2. Primary Outcome: Ankle Strength
Description: Ankle strength will be measured in response to the average of three 5-second dorsiflexion maximum voluntary isometric contractions per 30 seconds of relaxation in-between using a dynamometer (RoMech Digital Hanging Scale).
Time Frame: an average of 4 weeks (phase II).
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Active E-Stim | Electrical Stimulation - Sham
Number analyzed (Participants) | 10 | 8
Kg | 8.5 (4.2) | 7.9 (3.7)

3. Secondary Outcome: Plantar Oxyhemoglobin
Description: Percentage of oxyhemoglobin (OxyHb) will be measured using a validated near-infrared (NIR) camera (Snapshot NIR, KENT Imaging Inc., Calgary, AB, Can) that detects an approximate value of real-time OxyHb level in superficial tissue. The metatarsus area including the five toes will be traced. Data reported includes plantar oxyhemoglobin after 10 minutes of stopping 1 hour of electrical stimulation therapy.
Time Frame: an average of 4 weeks (phase II)
Measure: Mean (Standard Deviation); unit: Percentage of oxyhemoglobin
Arm/Group | Active E-Stim | Electrical Stimulation - Sham
Number analyzed (Participants) | 10 | 8
Percentage of oxyhemoglobin | .57 (.07) | .54 (.06)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Active E-Stim | Electrical Stimulation - Sham
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT05198466/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT05198466/ICF_001.pdf